CLINICAL TRIAL: NCT03291080
Title: Relative Bioavailability and Comparative Pharmacokinetics of 13-CRA Oral Liquid and Extracted Capsule Formulations: a Randomised, Open Label, Multi-dose, Cross-over Clinical Trial in Patients Requiring Treatment Cycles of 13-CRA.
Brief Title: Oral Liquid 13-cis-retinoic Acid (13-CRA)
Acronym: My-CRA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INV500
Record Dates: First submitted 2017-07-19; First posted 2017-09-25 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid (Experimental): Oral liquid formulation of 13-Cis Retinoic Acid - test product.
  Interventions: Drug: Liquid 13-Cis Retinoic Acid
- Capsule (Experimental): Isotretinoin capsules (13-CRA extracted per standard of care)- reference product.
  Interventions: Drug: Extracted capsules 13-CRA

INTERVENTIONS:
Drug: Liquid 13-Cis Retinoic Acid — Liquid 13-Cis Retinoic Acid
  Other Names: Isotretinoin
  Arms: Liquid
Drug: Extracted capsules 13-CRA — Extracted capsules 13-CRA
  Other Names: Isotretinoin
  Arms: Capsule

SUMMARY:
An open label, randomised, multiple dose, cross-over relative bioavailability and pharmacokinetics trial of a novel oral liquid and capsule formulations of 13-CRA administered to patients from 0 months - < 21 years.

DETAILED DESCRIPTION:
All patients requiring at least two cycles of 13-CRA therapy will be eligible for recruitment into the trial.

13-CRA will be prescribed to patients according to local treatment protocols at each clinical site. The dose administered will be 200mg/m2/day for both test and reference product. Patients with a body weight of ≤12kg will receive a dose of 160 mg/m2/day.

The pharmacokinetics of 13-CRA liquid (test product) and extracted from capsule (reference product) will be evaluated over two months. Prior to the initiation of 13-CRA treatment as part of the trial, patients will be randomised to receive either liquid or capsule formulation in "My-CRA month 1". The patients will then cross-over to the alternative formulation in "My-CRA month 2". The patients on the trial who require further treatment will revert to standard therapy i.e. 13-CRA extracted from capsules according to local practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged from 0 years to < 21 years of age.
2. Patient with high risk neuroblastoma, or unresectable, unfavourable histology intermediate risk neuroblastoma the latter age ≥ 18 months at diagnosis
3. Patient who is scheduled to receive at least two treatment cycles of 13-CRA.
4. Patient who cannot swallow 13-CRA capsules (i.e. requires extraction of 13-CRA from the capsules).
5. Negative pregnancy test for females of child-bearing potential before initiation of treatment, and sexually active patients and partners agreeing to undertake adequate contraceptive measures (see section 4.5).
6. Provision of a single or double lumen central venous catheter for sampling (i.e. already in place).
7. Parent(s)/legal guardian able and willing to provide written informed consent for the patient to take part in the trial.
8. Where applicable, the patient should assent to undergo blood sampling for pharmacokinetic purposes and to allow physiological measurements to be made.

Exclusion Criteria:

1. Any clinically significant medical condition or abnormality, which, in the opinion of the investigator, might compromise the safety of the patient or which might interfere with the trial.
2. Diagnosis of high-risk neuroblastoma (HRNBL) which is currently being treated on the SIOPEN HRNBL trial (patients who have exited this trial will be eligible).
3. Known allergy to 13-CRA or any of the excipients.
4. Inadequate contraception measures in females of childbearing age.
5. Receiving concomitant treatment with tetracyclines.

Prior to each cycle:

1. Total bilirubin ≤ 1.5 x normal, and (SGPT) ALT ≤ 5 x normal. Veno-occlusive disease if present, should be stable or improving.
2. Skin toxicity no greater than CTCAE Grade 1(10)
3. Serum triglycerides <5.65mmol/L.
4. No haematuria and / or proteinuria on urinalysis.
5. Serum calcium ≤ 2.9mmol/L.
6. Serum creatinine based on age / gender as follows:

   Age Maximum Serum Creatinine µmol/L Male Female 1 month to < 6 months 35 35 6 months to < 1 year 44 44 1 to < 2 years 53 53 2 to < 6 years 70 70 6 to < 10 years 88 88 10 to < 13 years 106 106 13 to < 16 years 132 124

   ≥ 16 years 150 124
7. Patients with a seizure disorder must be well controlled and taking anticonvulsants. CNS toxicity < grade 2 (CTCAE).

Withdrawal Criteria:

1. Positive pregnancy test - pregnancy testing will be undertaken before treatment commences and routinely before each course of treatment in females of childbearing potential. If a patient is found to be pregnant during the trial, the next course of treatment will not be given until the pregnancy has been discussed with the treating clinician, and the patient will be withdrawn from the trial whether or not treatment is continued.
2. Request of the patient, for any reason.
3. Discretion of the investigator.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussain Mulla, PhD, Study Director — Nova Laboratories Limited
Locations (10):
- United Kingdom (10):
  - Bruce Morland, Birmingham
  - Dr Antony Ng, Bristol
  - Dr Amos Burke, Cambridge
  - Mark Brougham, Edinburgh
  - Dr Martin Elliott, Leeds
  - Dr Guiseppe Barone, London
  - Dr Guy Makin, Manchester
  - Dr Madhumita Dandapani, Nottingham
  - Kate Wheeler, Oxford
  - Sucheta Vaidya, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veal GJ, Tweddle DA, Visser J, Errington J, Buck H, Marange J, Moss J, Joseph S, Mulla H. Pharmacokinetics and Safety of a Novel Oral Liquid Formulation of 13-cis Retinoic Acid in Children with Neuroblastoma: A Randomized Crossover Clinical Trial. Cancers (Basel). 2021 Apr 14;13(8):1868. doi: 10.3390/cancers13081868. PMID 33919763

RESULTS

PARTICIPANT FLOW:
Groups:
- First Oral Liquid, Then Capsule: Oral liquid formulation of 13-Cis Retinoic Acid (test product) in the first cycle. Then extracted 13-CRA capsule (reference product) in the second cycle.
- First Capsule, Then Oral Liquid: 13-CRA capsules extracted per standard of care (reference product) in the first cycle. Then oral liquid formulation of 13-CRA (test product) in the second cycle.
Period: First Cycle (2 Weeks)
Arm/Group | First Oral Liquid, Then Capsule | First Capsule, Then Oral Liquid
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | First Oral Liquid, Then Capsule | First Capsule, Then Oral Liquid
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Second Cylcle (2 Weeks)
Arm/Group | First Oral Liquid, Then Capsule | First Capsule, Then Oral Liquid
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Liquid First: Oral liquid formulation of 13-Cis Retinoic Acid (test product) administered in Cycle 1, then 13-CRA extracted capsules (reference product) administered in Cycle 2. The daily dose in each cycle was 200mg per m^2 (in 2 divided doses), reduced to 160 mg per m^2 if weight < 12 kg
- Extracted Capsule First: 13-CRA extracted capsules (reference product) administered in Cycle 1, then oral liquid formulation of 13-Cis Retinoic Acid (test product) administered in Cycle 2. The daily dose in each cycle was 200mg per m^2 (in 2 divided doses), reduced to 160 mg per m^2 if weight < 12 kg
- Total: Total of all reporting groups
Arm/Group | Liquid First | Extracted Capsule First | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 9 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 8 | 7 | 15
  Race: Asian or Asian British | 2 | 2 | 4
  Race: Other | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: Metre] | 0.974 (0.113) | 1.062 (0.21) | 1.009 (0.163)
Weight [Mean (Standard Deviation); unit: Kg] | 14.66 (3.47) | 18.96 (9.09) | 16.3 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability
Description: Relative bioavailability (Area under the curve) of 13-CRA administered as oral liquid (test) and extracted capsule (reference) formulations.
Time Frame: On day 1 and 14 of treatment
Population: Relative bioavailability - AUC (h.ng/mL)
Measure: Mean (Standard Deviation); unit: (h.ng/mL)
Groups:
- 13-CRA Oral Liquid: Oral liquid formulation - test product
- 13-CRA Extracted Capsule: Oral liquid formulation - reference product
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(h.ng/mL) | 10009.0 (3672.97) | 6075.9 (2090.66)

2. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetic parameter for 13 CRA extracted capsules versus oral liquid formulation
Time Frame: On day 1 and 14 of treatment
Measure: Mean (Standard Deviation); unit: (ng/mL)
Groups:
- 13-CRA Extracted Capsule: Extracted Capsules- reference product
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(ng/mL) | 1237.6 (662.67) | 748.2 (379.28)

3. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Pharmacokinetic parameter for 13 CRA extracted capsules versus oral liquid formulation
Time Frame: On day 1 and 14 of treatment
Measure: Mean (Standard Deviation); unit: (h)
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(h) | 3.2 (0.76) | 3.0 (0.76)

4. Secondary Outcome: Area Under Plasma Concentration Time Curve (AUC) Metabolite
Description: Pharmacokinetic parameter for 13 CRA extracted capsules versus oral liquid formulation- metabolite 4-oxo-13-cisRA
Time Frame: On day 1 and 14 of treatment
Measure: Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(h*ng/mL) | 38462.3 (18913.60) | 23312.7 (10947.59)

5. Secondary Outcome: Cmax (ng/mL)- Metabolite
Description: Pharmacokinetic parameter for metabolite 4-oxo-13-cisRA PK
Time Frame: On day 1 and 14 of treatment
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(ng/mL) | 3366.2 (1648.08) | 2039.1 (952.23)

6. Secondary Outcome: T Max of Metabolite
Description: T max for metabolite -4-oxo-13-cisRA PK
Time Frame: On day 1 and 14 of treatment
Measure: Mean (Standard Deviation); unit: (h)
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
Number analyzed (Participants) | 20 | 20
(h) | 7.1 (1.16) | 6.9 (1.16)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 months.
Arm/Group | 13-CRA Oral Liquid | 13-CRA Extracted Capsule
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 10/20 | 5/20
Other Adverse Events (participants affected / at risk) | 18/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13-CRA Oral Liquid (N=20) | 13-CRA Extracted Capsule (N=20)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 2 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncitial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Enteric neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13-CRA Oral Liquid (N=20) | 13-CRA Extracted Capsule (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Chapped Lips (Gastrointestinal disorders) | 8 (9) | 6 (6)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 5 (6)
Vomiting (Gastrointestinal disorders) | 3 (5) | 4 (5)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 6 (8)
Swelling face (General disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (12)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03291080/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03291080/SAP_001.pdf